CLINICAL TRIAL: NCT02053623
Title: Evaluation of a Novel Non-Invasive Electrocardiogram-Assisted Blood Pressure Monitor Against Invasive Intra-Arterial Pressure Monitoring - A Pilot Study
Brief Title: Evaluation of a Non-Invasive Electrocardiogram-Assisted Blood Pressure Monitor
Status: Terminated | Type: Observational
Why Stopped: Technical issues & lack of funds
Sponsor: Health Parametrics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HPI-219939
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypertension; Atrial Fibrillation; Obesity; Heart Failure; Atherosclerosis
MeSH Terms: conditions — Hypertension; Atrial Fibrillation; Obesity; Heart Failure; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Approximately one billion people suffer from hypertension worldwide. At least 10% of this population, that is, 100 million people, also suffers from associated chronic conditions namely, atrial fibrillation (AF), obesity, arterial stiffness (AS), and heart failure (HF). Personal interaction with medical practitioners (doctors) and review of published clinical research confirms that current non-invasive automatic blood pressure (BP) monitors that rely on BP pulse analysis alone cannot provide accurate measurement due to the unpredictable/weak nature of BP pulses in the above-mentioned chronic conditions. Lack of accuracy in BP estimation can lead to wrong diagnoses and hence to complications such as stokes and heart attacks.

The Sponsor is developing a novel non-invasive BP monitor that is similar to existing automatic monitors yet is capable of acquiring and analyzing electrocardiogram (ECG) data in conjunction with BP pulse data to provide better and more accurate measurements in the above chronic conditions.

The objective of this clinical trial is to evaluate the performance of this ECG-assisted BP monitor against invasive BP measurements in a small group of patients who suffer from the above conditions.

ELIGIBILITY:
Inclusion:

1. Patients undergoing an angiography in the catheterization lab who also suffer from at least one of the following chronic conditions:

   * Established diagnosis of AF.
   * Obesity characterized by a BMI > 40 (extremely high, Class III).
   * Established diagnosis of AS.
   * Established diagnosis of HF.
2. Age ≥ 18 years.

Exclusion:

1. Patients unwilling or unable to comply with study requirements.
2. Failure to sign the informed consent form.
3. Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit a minimum of 20 qualified adult patients who come to the catheterization lab at the University of Ottawa Heart Institute for an angiography. The patients will have at least one of the following chronic conditions: atrial fibrillation, obesity, atherosclerosis, and heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2015-05-21 (Actual); Study Completion 2015-07-02 (Actual)

PRIMARY OUTCOMES:
Accurate and Consistent Blood Pressure Measurement | 12 months
  We expect to demonstrate that our automated non-invasive ECG-assisted BP monitoring technology can provide accurate and consistent diastolic & systolic pressure measurements in chronic patient conditions (namely AF, obesity, AS, and HF) in which current non-invasive oscillometric technologies tend to be unreliable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada